CLINICAL TRIAL: NCT06089928
Title: Fixation Free Sandwich Osteotomy for Vertical Ridge Augmentation in Aesthetic Zone Versus Conventional Sandwich Osteotomy: A Randomized Controlled Clinical Trial
Brief Title: Fixation Free Sandwich Osteotomy With an Interpositional Inlay Graft in Compere to Conventional Sandwich Osteotomy
Acronym: sandwich
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ashour Ammar, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: segmental osteotomy
Record Dates: First submitted 2023-10-10; First posted 2023-10-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Vertical Ridge Deficiency; Atrophic Maxilla
Keywords: sandwich osteotomy; vertical augmentation,; aesthetic zone; Interpositional graft; fixation free
MeSH Terms: conditions — Atrophic Maxilla

STUDY DESIGN:
Intervention Model Description: clinical and radiographical comparisons of newly formed bone following vertical ridge augmentation which is achieved by use sandwich osteotomy with Interpositional inlay graft (ramus block) without fixation (test group), and same procedure with using micro-plates and screws as a mean of fixation (control group).
Who Masked: Participant, Outcomes Assessor
Masking Description: both the participant and outcome assessor would not know to which group of study they belong investigator can not be masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fixation free (Active Comparator): sandwich osteotomy with Interpositional graft without fixation.
  Interventions: Procedure: vertical augmentation
- conventional sandwich osteotomy (Active Comparator): sandwich osteotomy with Interpositional graft with fixation.
  Interventions: Procedure: vertical augmentation

INTERVENTIONS:
Procedure: vertical augmentation — sandwich osteotomy with an Interpositional inlay graft
  Other Names: segmental osteotomy with Interpositional graft

SUMMARY:
The atrophatic anterior maxilla present a considerable challenge for both surgical and prosthetic rehabilitation, as it may require bone augmentation to enable implant placement. The techniques proposed for vertical augmentation of the alveolar ridge include distraction osteogenesis, only grafting, and sandwich osteoplasty. Sandwich osteotomy is reported to provide more stable and predictable results with respect to the height of the alveolar ridge. The main advantage of osteotomy techniques that employ Interpositional bone grafts is reported to be the improved blood supply in the augmented region.

DETAILED DESCRIPTION:
the investigators aim to evaluate the radiographical, clinical differences of newly formed bone following vertical maxillary ridge augmentation using sandwich inlay with autogenous bone block from the rums without fixation (study group I) compared to same procedure with fixation (micro plates and screw) (control group).

description of intervention:

1) diagnostic procedure:

* All Participant will be selected according to inclusion and exclusion criteria.
* Comprehensive clinical examination and understanding of patient's chief complaints will be carried out.
* All participants will be informed about the surgical treatment procedure and will provide their written consent to participate in the study.
* Preoperative panoramic radiograph will be requested prior as general screening for any pathosis and primary maxillary anterior residual bone height assessment.
* A (CBCT) scan will be requested for each patient to confirm amount of horizontal and vertical bone, to exactly measure the amount of bone height and to plan and guide surgical procedures of block graft.
* Alginate Impressions of upper & lower jaws will be taken for acquiring diagnostic dental casts.

intra-surgical procedure :

Harvesting procedures of the mandibular ramus block graft:

After administering local anesthesia, a soft tissue incision will be made in the posterior mandible to create an envelope flap similar to that created in a third molar extraction, with an external oblique incision extending anteriorly into the buccal sulcus of the respective molar sites. A mucoperiosteal full-thickness flap will be then reflected with a sharp periosteal elevator, exposing the lateral aspect of the ramus. Osteotomies to take ABB will be performed in the ramus using trephine drills. The size of the block depended on the size of the graft needed. The size of the graft will be adjected with diamond discs under saline irrigation. Donor sites will be closed after the bone graft procedure will be completed. Recipient site preparation:

Following the administration of local anesthesia, a soft tissue incision will be performed. After a full-thickness mucoperiosteal flap will be reflected, the alveolar bone exposed. The edentulous area and the residual bone ridge will be prepared carefully to receive the bone graft; the defect dimensions will be measured with a periodontal probe to determine the approximate size of the block graft to be harvested or amount of particle bone graft needed.

Three full-thickness bony cuts will be performed. Two vertical stop cuts will be made using a tungsten carbide disc at the distal ends of the mid-crestal bony cut on the facial surface of alveolar ridge; the vertical cuts will be 3 mm from the neighboring teeth. The above-described cuts will be revised using ridge-splitting osteotomes (fine chisels) of sequential width (2 mm, 3 mm) and a lightweight mallet. The rectangular bony segment (transport segment) will be mobilized occlusally and be pedicled on the palatal mucoperiosteum. The autogenous blocks will be fitted between the mobilized segment and the basal bone, and the remining gap will be filled with particulated autogenous bone, in test group; there is no mean of fixation will be used while in the control group the segment will be fixed using micro-plates and screws. Scoring will be done to allow tension-free closure.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Adulte patient (18-60 y.)
* Highly motivated patient with good oral hygiene
* No systematic diseases or conditions known to alter bone healing.
* No local pathosis that may interfere with bone healing.
* No recent history of augmentation procedure at the same area.
* Criteria of the edentulous ridge:
* The anterior maxillary vertical dimension is minimum 10mm, measured from the crest of the ridge to the nasal floor.
* Horizontal ridge dimension remains normal; at least 6mm.
* The minimum number of the missing teeth is minimum 2 teeth and the maximum will be the six anteriors.
* There will be increased inter-arch space compared with the adjacent teeth.

Exclusion Criteria:

* uncontrolled Diabetes mellitus (DM)
* pregnancy
* uncontrolled local factors(periodontitis), or acute infection related to the aera.
* smoking: more than 20 cigarettes \day
* intravenous bisphosphonate
* patients who had received radiation treatment in the head and neck region.
* previous bone augmentation in the site within 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
radiographical bone gain | 4-months
  amount of vertical bone gain in millimeter using cone beam CT scan
radiographical bone change | 4- months
  amount of bone change in millimeter using cone beam CT scan

SECONDARY OUTCOMES:
clinical pain | 1-3days
  pain measure on a scale using visual analog scale
clinical edema | 1-7 days
  measure by edema index in terms of grades with minimum 1(better outcome and maximum 4( worse outcome)
clinical infection | 1-5 days
  binary as present or not present
clinical dehiscence | 1-30 days
  binary as present or not present

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected individual participant data including diagnosis, treatment plane, surgical intervention, outcome assessment, results will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 4-months follow-up
Access Criteria: open